CLINICAL TRIAL: NCT06295731
Title: A Phase 2/3, Randomized Study of INBRX-106 Combined With Pembrolizumab Versus Pembrolizumab as First Line Treatment for Patients With Recurrent or Metastatic (R/M) Head and Neck Squamous Cell Carcinoma (HNSCC) Expressing PD-L1 (CPS ≥20) (HexAgon-HN)
Brief Title: INBRX-106 in Combination With Pembrolizumab in First-line PD-L1 CPS≥20 HNSCC
Acronym: HexAgon-HN
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Inhibrx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INBRX106-01-201; EU CT (Other: 2024-515538-34)
Record Dates: First submitted 2024-02-22; First posted 2024-03-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: OX40 receptor agonist; PD-L1 positive; Pembrolizumab; Immunotherapy; Chemotherapy-free; HNSCC; Head and Neck Cancer; Keytruda; Oropharyngeal cancer; Hypopharyngeal cancer; Laryngeal cancer; Oral cancer; INBRX-106
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 2: open label; Phase 3: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INBRX-106 plus pembrolizumab (Experimental): Participants will receive INBRX-106 plus pembrolizumab, both given by intravenous (IV) infusion every 3 weeks (QW3)
  Interventions: Drug: INBRX-106; Drug: Pembrolizumab
- pembrolizumab monotherapy (+ placebo in phase 3 part) (Active Comparator): Participants will receive pembrolizumab (plus placebo in Phase 3), given by intravenous (IV) infusion every 3 weeks (QW3)
  Interventions: Drug: INBRX-106; Drug: Pembrolizumab

INTERVENTIONS:
Drug: INBRX-106 — INBRX-106 by intravenous (IV) infusion, given every 3 weeks (QW3)
  Other Names: Hexavalent OX40 agonist antibody
Drug: Pembrolizumab — Pembrolizumab 200 mg by intravenous (IV) infusion, given every 3 weeks (QW3)
  Other Names: Keytruda

SUMMARY:
This seamless phase 2/3 randomized controlled study will evaluate the efficacy and safety of the hexavalent OX40 agonist antibody INBRX-106 combined with the anti-PD-1 antibody pembrolizumab versus pembrolizumab (+ placebo in phase 3) as first-line treatment for patients with locally advanced recurrent or metastatic head and neck squamous cell carcinoma (R/M HSNSCC) incurable by local therapies, expressing PD-L1 with a combined proportion score (CPS) ≥20.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of metastatic, recurrent head and neck squamous cell carcinoma (HNSCC) that is considered incurable by local therapies.
* Has tumor PD-L1 expression of CPS ≥20. Tumor tissue must be provided for PD-L1 biomarker analysis.
* Has human papilloma virus (HPV) testing results for oropharyngeal cancer by p16 immunohistochemistry (IHC) testing.
* Has measurable disease per RECIST 1.1 guidelines.
* Has the primary tumor location of the oral cavity, oropharynx, hypopharynx, or larynx.
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Female patients of childbearing potential must have a negative highly sensitive pregnancy test within 72 hours prior to randomization and must not be breastfeeding.
* Male and female patients of childbearing potential must be willing to completely abstain from heterosexual sex or agree to use a highly effective method of contraception.

Exclusion Criteria:

* Has primary tumor site (any histology) of nasopharynx or salivary glands or occult primary site.
* Has received prior systemic therapy (eg, prior chemo-, immune-, or biologic therapy) for locally advanced unresectable or metastatic HNSCC.

  * Prior systemic therapy completed >6 months prior to signing informed consent is allowed if given as part of multimodal treatment for locoregionally advanced disease with curative intent, and no PD/recurrence occurred within 6 months of its completion. Prior systemic immunotherapy in the locoregionally advanced disease with curative intent, including but not limited to anti-PD-(L)1 agents, is allowed if PD/recurrence occurred ≥12 months after its completion.
* Has clinically active central nervous system metastases and/or carcinomatous meningitis.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Rapidly progressing disease or with features that may confer a high risk of tumor-associated hemorrhage or uncontrolled tumor pain.
* Current or history of immune-related disease that required systemic treatment in past 2 years, except for replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Objective Response Rate (ORR) | up to 6 months
  ORR is defined as the proportion of patients with a complete response (CR) or partial response (PR) on 2 consecutive occasions ≥4 weeks apart, per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Phase 3: Progression-Free Survival (PFS) | From randomization to first occurrence of progressive disease (PD) or death (up to 4 years)
  PFS is defined as the time from randomization to first occurrence of PD, as determined by the Investigator according to RECIST v 1.1, or death from any cause (whichever occurs first).
Phase 3: Overall Survival (OS) | From randomization until death from any cause (up to 4 years)
  OS is the time from randomization to death due to any cause

SECONDARY OUTCOMES:
Phase 3: Objective Response Rate (ORR) | From randomization until treatment discontinuation (up to 2 years)
  ORR is defined as the proportion of patients with a CR or PR on 2 consecutive occasions ≥4 weeks apart, per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Duration of Response (DOR) | From the first occurrence of a documented objective response to PD or death (up to 4 years)
  DOR is defined as the time from the first occurrence of a documented objective response to PD, as determined by the Investigator according to RECIST v1.1, or death from any cause (whichever occurs first)
Clinical Benefit Rate (CBR) | From randomization until treatment discontinuation (up to 2 years)
  CBR is defined as the proportion of patients with stable disease (SD) for ≥12 weeks or a CR or PR, as determined by the Investigator according to RECIST v1.1.
Phase 3: Time to Chemotherapy (TTCtx) | From randomization until the start of chemotherapy or death (up to 4 years)
  TTCtx is defined as the time from randomization until the start date of chemotherapy or death from any cause (whichever occurs first).
Time to Confirmed Deterioration (TTCD) in Pain Presence and Interference | From randomization until treatment discontinuation (up to 2 years)
  TTCD in pain presence and interference is defined as the time from randomization to the first documentation of ≥10-point increase in pain score, as determined using the European Organization for Research and Treatment of Cancer Quality of Life-Core 30 (EORTC QLQ-C30) questionnaire
TTCD in physical functioning (PF) | From randomization until treatment discontinuation (up to 2 years)
  TTCD in PF is defined as the time from randomization to the first documentation of a ≥10 point decrease from baseline in the Quality of Life-Core 30 (EORTC QLQ-C30) linearly transformed PF scale score.
TTCD in role functioning (RF) | From randomization until treatment discontinuation (up to 2 years)
  TTCD in RF is defined as the time from randomization to the first documentation of a ≥10 point decrease from baseline in the Quality of Life-Core 30 (EORTC QLQ-C30) linearly transformed RF scale score.
TTCD in Global Health Status/quality of life (GHS/QoL) | From randomization until treatment discontinuation (up to 2 years)
  TTCD in GHS/QoL is defined as the time from randomization to the first documentation of a ≥10 point decrease from baseline in the Quality of Life-Core 30 (EORTC QLQ-C30) linearly transformed GHS/QoL scale score.
Incidence and severity of Adverse Events (AEs) | Up to approximately 24 months
  Incidence will be reported as the number of participants with at least one adverse event, with severity determined according to the National Cancer Institute Criteria for Adverse Events, version 5 (NCI CTCAE v 5.0)
Number of patients who experienced abnormalities in vital signs and clinical laboratory parameters | Up to approximately 24 months
  Vital signs include respiratory rate, pulse rate, systolic and diastolic blood pressure, and temperature. Clinical laboratory parameter include hematology and biochemistry tests over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Study Director — Inhibrx Biosciences, Inc
Locations (88):
- United States (26):
  - City of Hope Medical Center, Duarte, California
  - Los Angeles Cancer Network (LACN), Los Angeles, California
  - Sutter Health, Sacramento, California
  - UC Davis, Sacramento, California
  - Medical Oncology Associates of San Diego, San Diego, California
  - Sarcoma Oncology Center, Santa Monica, California
  - ChristianaCare Health Services, Newark, Delaware
  - University of Florida UF Health Cancer Center, Gainesville, Florida
  - The Oncology Institute of Hope & Innovation, Miami, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Cleveland Clinic Florida, The Maroone Cancer Center, Weston, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University St. Louis, St Louis, Missouri
  - Intermountain Health, St. Vincent Regional Hospital, Cancer Centers of Montana, Billings, Montana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Christus St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Oklahoma University Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - CHRISTUS Spohn Cancer Center, Corpus Christi, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Belgium (4):
  - Antwerp University Hospital, Edegem, Antwerp
  - University Hospital Brussels, Jette
  - Chu Ucl Namur Site De Sainte-Elisabeth, Namur
  - Vitaz, Sint-Niklaas
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment - "Uni Hospital" Ltd, Medical Oncology Dept, Panagyurishte
  - Complex Oncological Center Plovdiv EOOD Dept of Med Oncology and Oncological Diseases in Hematology, Plovdiv
  - Uni Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD Clinic of Medical Oncology, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Sofia, Department of Medical Oncology, Sofia
- France (5):
  - CH Annecy Genevois, Annecy, Epagny Metz Tessy
  - UNEOS-Hopital R.SCHUMAN, Metz, Moselle
  - Centre Jean Perrin, Clermont-Ferrand
  - Cenre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
- Italy (4):
  - Istituto Nazionale Tumori IRCCS - Fondazione Giovanni Pascale (National Cancer Institute), Napoli, Naples
  - Istituto Nazionale Tumori IRCCS - (National Cancer Institute), Milan
  - European Institute of Oncology, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Malaysia (6):
  - Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Hospital Canselor Tuanku Muhriz (HCTM) UKM, Cheras, Kuala Lumpur
  - Sarawak General Hospital, Kuching, Sarawak
  - Thomson Hospital Kota Damansara, Petaling Jaya, Selangor
  - Beacon Hospital, Petaling Jaya
  - Institut Kanser Negara, Putrajaya
- Poland (3):
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy Oddział w Gliwicach, Gliwice
  - Przychodnia Lekarska KOMED, Konin
  - Provita Profamilia, Piotrkow Trybunalski
- Romania (4):
  - Sc Oncolab Srl, Craiova, Dolj
  - Sc Centrul de Oncologie Sf Nectarie Srl, Craiova, Dolj
  - ARENSIA Clinic Oncology Institute Bucharest, Bucharest
  - Arensia Exploratory Medicine S.R.L in collaboration with "Prof. Dr. Ion Chiricuta" Oncology Institute, Cluj-Napoca, Cluj
- South Korea (8):
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Gachon University Gil Medical Center of Korea, Seoul, Incheon
  - Keimyung University Dongsan Hospital of Korea, Daegu
  - Korea Cancer Center Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (9):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago, A Coruña
  - Intituto Catalán de Oncología, Barcelona, Catalonia
  - IOB / Institute of Oncology, Hospital Quirónsalud Barcelona, Barcelona, Gracia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Gregorio Marañón, Madrid, Retiro
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia
- Taiwan (6):
  - Taipei Veterans General Hospital, Taipei, Beitou District / R.o.c.
  - Taichung Veterans General Hospital, Taichung, China
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (8):
  - The Royal Marsden NHS Foundation Trust, Chelsea, Chelsea, London
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Northern Centre for Cancer Care, Freeman Hospital, Newcastle upon Tyne, Northumbria
  - The Royal Marsden NHS Foundation Trust, Sutton, Sutton, Surrey
  - NHS Grampian / Aberdeen Royal Infirmary, Aberdeen
  - Addenbrooke's Hospital, Cambridge
  - The Christie NHS Foundation Trust, Manchester
  - Norwich and Norfolk University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No